CLINICAL TRIAL: NCT04809545
Title: Evaluation of Personalized Soundscape Effects on Persons With Dementia; a Pilot Randomized Clinical Trial
Brief Title: Effect of Soundscape on People With Dementia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: University Ghent (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20-5067
Record Dates: First submitted 2021-03-17; First posted 2021-03-22 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Dementia; Behavioural and Psychiatric Symptoms of Dementia
Keywords: Soundscape; Sonic environment; Neuropsychiatric symptoms; Dementia; Environmental design
MeSH Terms: conditions — Dementia | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Single blind repeated-measures randomized controlled study with two parallel arms, Intervention and Treatment As Usual (TAU) with a 2:4:1 design (two baseline measures, four intervention measures, 1 post-intervention)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single-blind study where the intervention is delivered outside of the hours of the investigator and outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The study intervention consists of the delivery of a soundscape in the private rooms of the participant during the morning and evening. The soundscape is personalized and consists of a collection of natural sounds, birdsongs, kitchen sounds, music, bell sound, outdoor sounds, water/rain sounds, and similar.
  Interventions: Other: Acusticare
- Treatment as Usual (Active Comparator): As part of usual care, patients on the Specialized Dementia Unit receive a comprehensive assessment of their health and symptoms of dementia involving consultation by a geriatric psychiatrist, geriatrician, physical therapist, occupational therapist, and recreation therapist, and pharmacological and non-pharmacological treatment plans are developed and executed. All participants in the study will receive this standard of care
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Acusticare — Acusticare is an internet connected speaker which delivers an environmental intervention by playing sounds to adjust the soundscape in the room.
  Arms: Intervention
Other: Treatment as usual — Usual care provided on the Specialized Dementia Unit
  Arms: Treatment as Usual

SUMMARY:
In the last few decades, insights into the impact of the sonic environment on persons have grown to include not only the adverse effects of extensive mechanical noise but also the beneficial effects of a well-designed sonic environment. People with dementia, however, perceive and understand the sonic environment differently. The most obvious difference is that the meanings they may give to the sounds they notice due to changing mental associations. However, also at an earlier perceptual stage, attention focusing and gating may be affected, reducing their ability to analyze a complex auditory scene. Behaviour associated with the appraisal of the sound environment may change with the emergence of dementia.

The objective of this study is to determine the effect size of a carefully tuned personalized sonic environment (delivered via AcustiCare) on agitation and distress (NPI and PAS), night sleep and stress (Via wristband) and on quality of life (QUALIDEM) in a population of older adults with dementia and behavioural symptoms.

DETAILED DESCRIPTION:
Research has shown the positive effect of natural and non-natural soundscape on people with severe or profound intellectual disabilities (Andringa & van den Bosch, 2013). Sound plays a role in generating a feeling of safety, in influencing the mood, and triggering a specific action. Bringing sound with this purpose, as targeted to the current activity can improve the behaviour. There is substantial research on the effect of noise (unwanted sound) on people's health and well-being. The health outcomes vary, but include cardiovascular disease, sleep disturbance, and annoyance.

In a previous study in people with dementia by the Belgian investigators in this study (Devos et al., 2019), they observed positive staff outcome measures, reflecting the value of the soundscape in improving their ability to provide care to people with dementia. They did not directly assess the benefits to residents in that study. There were no harms documented in the study, and if residents reacted not well to specific sound, the sound was removed from the soundscape.

The aim of this study is to build upon the previous research and evaluate the effect of a personalized soundscape on the well-being and behaviour of persons with dementia. In the soundscapes, we use only recognizable sounds, sounds that give persons with dementia a feeling of 'safety' or sounds that focus on the orientation (in time, place). We try to add a recognizable (safe, orientating) sound through the soundscape system. This soundscape supports the environment and makes the environment feel safer and more 'clear' for residents with dementia. In the previous research through co-design process with staff and family member the sounds were chosen (Devos et al, 2018).

Most of the existing studies in the field of the acoustic environment in health care are descriptive, and there is a need for a more rigorous evaluation of interventions. By using a pilot Randomized Control Trial (RCT) design, we will be able to establish the effect size of soundscape on outcomes of interest in this population of people with dementia. These results will support evidence-based practices by healthcare providers, architects, engineers and designers in implementing environmental health factors and designing better care facilities for people with dementia in the future.

The objective of this study is thus to determine the effect size of a carefully tuned personalized sonic environment (delivered via AcustiCare) on agitation and distress (NPI and PAS), night sleep and stress (Via wristband) and on quality of life (QUALIDEM).

ELIGIBILITY:
Inclusion Criteria:

1. 65 years or older
2. Diagnosis of Dementia
3. Symptoms of BPSD at baseline
4. English speaking
5. Assigned a private room with AcustiCare installed

Exclusion Criteria:

1. Severe hearing impairment
2. Receiving end-of-life care

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change over 6 weeks in Neuropsychiatric Inventory- total score | Baseline and weekly over 6 weeks
  Assessments of behavioural and psychological symptoms of dementia on a weekly basis over the study duration will be included in a longitudinal mixed effects model as part of a repeated measures design

SECONDARY OUTCOMES:
Change over 6 weeks in the Pittsburgh Agitation Scale-- Resisting Care subscale | Baseline and weekly over 6 weeks
  Assessment of resistance to care on a weekly basis over the study duration will be included in a longitudinal mixed effects model as part of a repeated measures design
Change over 6 weeks in the Pittsburgh Agitation Scale-- Total score | Baseline and weekly over 6 weeks
  Assessment of behavioural symptoms on a weekly basis over the study duration will be included in a longitudinal mixed effects model as part of a repeated measures design
Change over 6 weeks in Neuropsychiatric Inventory Agitation Subscale | Baseline and weekly over 6 weeks
  Assessment of agitation on a weekly basis over the study duration will be included in a longitudinal mixed effects model as part of a repeated measures design
Change over 6 weeks in Neuropsychiatric Inventory Aggression subscale | Baseline and weekly over 6 weeks
  Assessment of aggression on a weekly basis over the study duration will be included in a longitudinal mixed effects model as part of a repeated measures design
Change over 6 weeks in Neuropsychiatric Inventory Dysphoria subscale | Baseline and weekly over 6 weeks
  Assessment of dysphoria on a weekly basis over the study duration will be included in a longitudinal mixed effects model as part of a repeated measures design
Change in Neuropsychiatric Inventory Anxiety subscale | Baseline and weekly over 6 weeks
  Assessment of anxiety on a weekly basis over the study duration will be included in a longitudinal mixed effects model as part of a repeated measures design
Change in Qualidem | Baseline, Week 6
  Dementia-related quality of life

OTHER OUTCOMES:
Change in staff feedback on 5-point scale over 6 weeks | Baseline and daily over 6 weeks
  Staff can provide real-time feedback on a daily basis on resident mood and behaviour using a 5-button scale
Change in accelerometer-measured nocturnal activity level over time | Weeks 2,4,5 and 6
  Using an accelerometer, will assess activity levels overnight as a measure of sleep fragmentation
Change in heart rate variability over time | Weeks 2,4,5 and 6
  Heart rate variability as a measure of stress

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Iaboni, MD DPhil, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Rehabilitation Institute, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Devos P, Aletta F, Thomas P, Petrovic M, Vander Mynsbrugge T, Van de Velde D, De Vriendt P, Botteldooren D. Designing Supportive Soundscapes for Nursing Home Residents with Dementia. Int J Environ Res Public Health. 2019 Dec 4;16(24):4904. doi: 10.3390/ijerph16244904. PMID 31817300
- [Background] Devos, P., Aletta, F., Vander Mynsbrugge, T., Thomas, P., Filipan, K., Petrovic, M., ... & Botteldooren, D. (2018, December). Soundscape design for management of behavioral disorders: a pilot study among nursing home residents with dementia. In INTER-NOISE and NOISE-CON Congress and Conference Proceedings (Vol. 258, No. 5, pp. 2104-2111). Institute of Noise Control Engineerin
- [Derived] Talebzadeh A, Botteldooren D, Thomas P, Stewart S, Van de Velde D, De Vriendt P, Devos P, Iaboni A. Effect of Soundscape Augmentation on Behavioral Symptoms in People With Dementia: A Pilot Randomized Controlled Trial. Innov Aging. 2024 Aug 5;8(9):igae069. doi: 10.1093/geroni/igae069. eCollection 2024. PMID 39350940